CLINICAL TRIAL: NCT02966899
Title: Reversal of Right Ventricular Steatosis in Pulmonary Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never initiated
Sponsor: Wen-Chih Wu (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Wen-Chih Wu, Chief of Medical, Providence VA Medical Center
Organization: Providence VA Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 312231
Record Dates: First submitted 2016-11-11; First posted 2016-11-17 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary; Hypertension; Steatosis; Right Ventricular Failure
MeSH Terms: conditions — Hypertension, Pulmonary; Fatty Liver; Heart Failure | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 fatty acids (Experimental): 30 patients with pulmonary hypertension who are identified as having elevated myocardial triglyceride content by cardiac MRI will receive 4 grams/day of omega-3 fatty acids for six months.
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids

SUMMARY:
The goal of this study is to elucidate the relationship between myocardial right ventricular triglyceride content (steatosis) and right ventricular dysfunction in participants with pulmonary hypertension, and investigate reversibility of this phenotype with omega-3 fatty acid treatment.

DETAILED DESCRIPTION:
The investigators propose to treat 30 participants that are identified as having elevated myocardial triglyceride content (defined as greater than 0.50%) on cardiac MRI with 4 grams of omega-3 fatty acids daily for six months with a primary end point of reducing right ventricular steatosis and a secondary endpoint of improving RV systolic function. The investigators hypothesize that right ventricular steatosis by cardiac MRI will be associated with the degree of right ventricular systolic function by cardiac MRI. In the subset of participants with elevated baseline steatosis who are treated with a lipoprotective strategy, the investigators hypothesize that six months of therapy with omega-3 fatty acids will reduce myocardial steatosis and improve right ventricular systolic function.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women > 30 years of age with a diagnosis of pulmonary hypertension (defined as mean pulmonary arterial pressure ≥25 mmHg at rest on right heart catheterization)

Exclusion Criteria:

* Contraindication to MRI (e.g., metallic hazards or allergy to gadolinium)
* Renal dysfunction (eGFR < 60 ml/min/1.73m2 as estimated by the Modified Diet in Renal Disease formula)
* High risk features for nephrogenic systemic fibrosis (solitary kidney or prior renal transplant)
* Active pregnancy or breastfeeding (determined by urinary pregnancy test before CMR)
* Weight > 550 lb or waist diameter > 70 cm (limits for our Siemens Verio CMR system)
* Fish Allergy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Right ventricular myocardial triglyceride content (by cardiac MRI) in 30 participants with pulmonary hypertension | 6 months

SECONDARY OUTCOMES:
Right ventricular ejection fraction (by cardiac MRI) in 30 participants with pulmonary hypertension | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided